CLINICAL TRIAL: NCT00735995
Title: Effectiveness of Group and Individual Treatment of Childhood Anxiety Disorders in Community Clinics. A Randomized Controlled Trial.
Brief Title: Effectiveness of Cognitive Behavioral Therapy (CBT) for Child Anxiety Disorders in Community Clinics in Norway
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regionsenter for barn og unges psykiske helse (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Simon-Peter Neumer, dr. Simon-Peter Neumer, Regionsenter for barn og unges psykiske helse
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 186036/V50; 186036 (Other Grant/Funding Number: Norwegian Research Council)
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Separation Anxiety Disorder; Social Phobia; Generalized Anxiety Disorder
MeSH Terms: conditions — Anxiety, Separation; Phobia, Social; Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy; Population Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Individual CBT
  Interventions: Behavioral: Cognitive behavioral therapy (individual)
- B (Experimental): Group CBT
  Interventions: Behavioral: Cognitive behavioral therapy (group)
- C (No Intervention): Waiting-list control

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (individual) — The Coping Cat program, 12 weekly sessions, two additional parent meetings
  Arms: A
Behavioral: Cognitive behavioral therapy (group) — The Coping Cat program, 12 weekly sessions, two additional parent meetings
  Arms: B

SUMMARY:
The purpose of this study is to assess the effectiveness of a cognitive-behavioral intervention for children aged 7 to 12 years with anxiety disorders who are referred to ordinary community clinics. The treatment will be conducted as individual therapy or group therapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of separation anxiety disorder, social phobia or generalized anxiety disorder based on the ADIS interview schedule, DSM-IV criteria

Exclusion Criteria:

* Pervasive Developmental Disorder
* Psychotic symptoms
* Intelligence score < 70
* Use of medications with anxiety reducing effects during treatment
* Neither parent competent in Norwegian language

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2008-08; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Status of primary anxiety disorder at inclusion based on the ADIS interview schedule with parents and youth | post-treatment and 2 year follow-up

SECONDARY OUTCOMES:
Symptom score on the MASC | post-treatment and 2 year follow-up
CGAS | post-treatment and 2 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Simon-Peter Neumer, dr.philos, Principal Investigator — Regionsenter for barn og unges psykiske helse
Locations (3):
- Norway (3):
  - Akershus Universitetssykehus HF, Lorenskog
  - Sykehuset Asker og Baerum, Baerum BUP, Rud
  - Sykehus Telemark Helseforetak, Skien og Porsgrunn BUP, Skien

REFERENCES:
- [Result] Gere MK, Hagen KA, Villabo MA, Arnberg K, Neumer SP, Torgersen S. Fathers' mental health as a protective factor in the relationship between maternal and child depressive symptoms. Depress Anxiety. 2013 Jan;30(1):31-8. doi: 10.1002/da.22010. Epub 2012 Oct 25. PMID 23108976
- [Result] Villabo MA, Cummings CM, Gere MK, Torgersen S, Kendall PC. Anxious youth in research and service clinics. J Anxiety Disord. 2013 Jan;27(1):16-24. doi: 10.1016/j.janxdis.2012.09.003. Epub 2012 Sep 25. PMID 23257654
- [Result] Villabø MA, Gere MK, Torgersen S, Arnberg K, Neumer SP, Kendall PC. Anxious self-statements in clinic-referred US and Norwegian anxiety-disordered youth. Cognitive Therapy and Research 37(4): 840-850, 2013.
- [Result] Gere MK, Villabo MA, Torgersen S, Kendall PC. Overprotective parenting and child anxiety: the role of co-occurring child behavior problems. J Anxiety Disord. 2012 Aug;26(6):642-9. doi: 10.1016/j.janxdis.2012.04.003. Epub 2012 May 14. PMID 22659077
- [Result] Villabo M, Gere M, Torgersen S, March JS, Kendall PC. Diagnostic efficiency of the child and parent versions of the Multidimensional Anxiety Scale for Children. J Clin Child Adolesc Psychol. 2012;41(1):75-85. doi: 10.1080/15374416.2012.632350. PMID 22233247
- [Result] Villabo MA, Narayanan M, Compton SN, Kendall PC, Neumer SP. Cognitive-behavioral therapy for youth anxiety: An effectiveness evaluation in community practice. J Consult Clin Psychol. 2018 Sep;86(9):751-764. doi: 10.1037/ccp0000326. PMID 30138014